CLINICAL TRIAL: NCT03652207
Title: The Effects of Palatinose™ on Weight Management and Body Composition in Overweight and Obese Individuals
Brief Title: Effects of Palatinose™ on Weight Management and Body Composition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beneo-Institute (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Beneo_OBU_101108Final
Record Dates: First submitted 2018-08-27; First posted 2018-08-29 (Actual); Last update posted 2018-08-29 (Actual); Status verified 2018-08

CONDITIONS: Overweight and Obesity; Diet Modification; Body Weight
MeSH Terms: conditions — Overweight; Obesity; Body Weight | interventions — isomaltulose; Sucrose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sucrose (Placebo Comparator): Test products i.e. low-fat yogurt drink, fruits drink and sweetener sachet for cereals containing sucrose
  Interventions: Other: Sucrose
- Palatinose(TM) (Experimental): Test products i.e. low-fat yogurt drink, fruits drink and sweetener sachet for cereals containing isomaltulose (Palatinose™)
  Interventions: Other: isomaltulose (Palatinose(TM)

INTERVENTIONS:
Other: isomaltulose (Palatinose(TM) — isomaltulose containing food products, i.e. low-fat yogurt drink, fruits drink and sweetener sachet for cereals, consumed within an energy-reduced diet
  Arms: Palatinose(TM)
Other: Sucrose — sucrose containing food products, i.e. low-fat yogurt drink, fruits drink and sweetener sachet for cereals, consumed within an energy-reduced diet
  Arms: Sucrose

SUMMARY:
The study aims to assess body weight and body composition changes in overweight and obese persons consuming an energy-reduced diet containing foods with either sucrose or isomaltulose (Palatinose(TM)) over a period of 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Subject is healthy at the time of pre-examination
* Subject has a BMI of 25 - 35 kg/m² and motivated to lose weight
* Subject is aged 18 - 60 years at the time of pre-examination

Exclusion Criteria:

* Person suffers from an acute or chronic disease
* Person has known dietary restrictions or allergies to Foods
* Intake of medications which interfere with body composition, appetite, satiety or food intake

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2009-04-20 (Actual); Primary Completion 2010-06-30 (Actual); Study Completion 2010-06-30 (Actual)

PRIMARY OUTCOMES:
Body Weight Change | 12 weeks
  Body weight Change over a 12-week period

SECONDARY OUTCOMES:
Body fat percentage | 12 weeks
  Body fat percentage measured using the BodPod
postprandial respiratory quotient (RQ) | 120 minutes postprandial
  postprandial energy metabolism, i.e. respiratory quotient (RQ) and fat oxidation measured by indirect calorimetry
BMI | 12 weeks
  Body mass index (kg/m2)
Waist circumference | 12 weeks
  Waist circumference assessed using a measuring tape

CONTACTS AND LOCATIONS:
Locations (1):
- Oxford Brookes University, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Maresch CC, Petry SF, Theis S, Bosy-Westphal A, Linn T. Low Glycemic Index Prototype Isomaltulose-Update of Clinical Trials. Nutrients. 2017 Apr 13;9(4):381. doi: 10.3390/nu9040381. PMID 28406437